CLINICAL TRIAL: NCT02713100
Title: Self Reported Level of Agitation of Patients Presenting to an Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leslie Zun, MD (Other)
Collaborators: Teva Pharma (Industry)
Responsible Party: Sponsor-Investigator, Leslie Zun, MD, Chairman, Mt Sinai Hospital, Chicago
Organization: Mt Sinai Hospital, Chicago (Other)
Other Study IDs: 14-15
Record Dates: First submitted 2014-10-20; First posted 2016-03-18 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Psychiatric Issue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: level of agitation — psychological pain

SUMMARY:
In recent years, there has been an emphasis on assessing patient's pain on presentation to emergency departments. The Joint Commission mandates that all patients who present with pain must have a pain assessment performed and addressed early in their care. Most emergency departments are using a self-reported assessment of pain using a 1-10 scale of pain. This self-reported level of pain is used to determining appropriate treatment. The Joint Commission has only dealt with somatic pain and has not addressed psychological related pain.

Many authors have written on psychological pain. It is described as introspective experience of negative emotions such as anger, despair, fear, grief, shame, guilt, hopelessness, loneliness and loss. The assessment of psychological pain has been used to describe patients with depression and suicidal thoughts and behaviors.

Study Significance The significance of this study is to determine if patients can communicate the level of psychological pain using the level of agitation as a surrogate marker. Studies have demonstrated that the staff's assessment of a patient's level of agitation is not based on an agitation scale nor uses any patient self-assessment of their level of agitation. If a self-assessment of a patient's level of agitation can be determined early in their care in the emergency setting, a proactive approach to treatment can occur. Proactive agitation treatment has the potential of reducing a patient's agitation and increasing their level of comfort. This early intervention can reduce the progression of agitation and the risk of injury to patients, families and staff.

Hypothesis The study null hypothesis is that the self-rated agitation scale will not have a significant level of correlation with the other measures of agitation (Brief Agitation Measure, Positive And Negative Syndrome Scale and Agitation Calmness Evaluation Scale). The secondary null hypothesis is that there is no difference between the level of agitation and the level of psychological pain, assessed with the Psychological Pain Assessment.

DETAILED DESCRIPTION:
In recent years, there has been an emphasis on assessing the patient's pain when the patient presents to emergency departments. The Joint Commission mandates that all patients who present with pain must have a pain assessment performed and addressed early in their care. Most emergency departments are using a self-reported assessment of pain using a 1-10 scale of pain. This self-reported level of pain is used to determine appropriate treatment. The Joint Commission has only dealt with somatic pain and has not addressed psychological pain.

Psychological pain is described as the introspective experience of negative emotions such as anger, despair, fear, grief, shame, guilt, hopelessness, loneliness and loss. The assessment of psychological pain has been used to describe patients with depression and suicidal symptoms.

Some in the field of emergency psychiatry believe patients who are agitated are exhibiting psychological pain, which some argue is no different than somatic pain. However, the principle of somatic pain assessment and treatment has never been applied to the assessment and treatment of psychological pain. Addressing a patient's level of agitation could be used to reduce their agitation and thereby, reduce their psychological pain.

Psychiatric patients frequently present to emergency departments (ED) across the country. Many of these patients are agitated, necessitating treatment for their agitation in the ED. Agitation is thought to be one way a patient expresses psychological pain. If one could assess and treat a patient's agitation, one may be able to reduce psychological pain.

Patients may exhibit various levels of agitation from mild to severe. Patients may progress from one level to the next or stay in one level. Moderate and severely agitated patients are difficult to evaluate and usually need treatment for their agitation. Some of these patients may become violent and injure themselves, staff or others. It is essential to identify patients who might be in the mild to moderate stage in order to prevent progression to severe agitation. This identification can provide a mechanism to determine who needs immediate treatment in the ED.

The treatment for these agitated patients frequently includes physical restraint, chemical treatment and seclusion. In a review of 13 published studies of adults in a patient psychiatric setting, a range of 1.9% to 66% patients had a need for seclusion and restraint. Another study found an average of 2 restraints on 17% of patients in an acute medical unit. In psychiatric emergency rooms, the percent of patients restrained (20-25%) was significantly higher than in an inpatient facility (7-20%) [8-11]. It was found 25.2% of teaching hospitals restrained at least one patient per day. An average of 3.7% of all ED patients needed restraint and seclusion, or restraint alone.

Although not frequently used in the emergency setting, there are many tools used to assessment agitation in the acute care setting including Brief Agitation Tool, Positive and Negative Syndrome Scale-Excited Component, Agitation Calmness Evaluation Scale, Richard Agitation Sedation Scale, Overt Agitation Severity Scale, and Agitation Behavior Scale.

Only one of these tools, Brief Agitation Tool, has been used to obtain a self-reported measure of agitation. However, this tool has been used only on students and outpatients; not in the emergency setting. Also, the tool was used to correlate agitation to suicidal symptoms.

Tools to measure a patient's psychological pain are limited. These include the Psychological Pain Assessment Scale and the Psychological Pain Assessment. These tools have been used in the study of depression and suicidal symptoms. It has not been evaluated on ED patients presenting with agitation.

The purpose of this study is to apply the same principle of assessing somatic pain to psychological pain using the level of agitation as a surrogate marker. This study will compare a self-rated agitation scale to the other measures of agitation (Brief Agitation Tool, Positive and Negative Syndrome Scale-Excited Component, and Agitation Behavior Scale). An analysis of the data will provide information concerning the accuracy of a self-administered scale in assessing agitation. The secondary purpose will to determine the correlation of a measure of psychological pain (Psychological Pain Assessment) to level of agitation.

Study Significance The significance of this study is to determine if patients can communicate the level of psychological pain using the level of agitation as a surrogate marker. If a self-assessment of a patient's level of agitation can be determined early their care in the emergency setting, a proactive active approach to treatment can occur. Proactive agitation treatment has the potential of reducing a patient's agitation and increasing their level of comfort. This early intervention can reduce the progression of agitation and the risk of injury to patients, families and staff.

Hypothesis The study null hypothesis is that the self-rated agitation scale will not have a significant level of correlation with the other measures of agitation. The secondary null hypothesis is that there is no difference between the level of agitation and the level of psychological pain.

Methods The study is a prospective enrollment with use of medical records & convenience sample of patients who present to the ED with a psychiatric complaint to determine their level of agitation and psychological pain. This study will be performed in a community, inner city teaching hospital ED with 55,000 visits per year. The city's police department has designated the hospital as the referral site for psychiatric patients in the southwest side of the city.

All patients will be evaluated by the emergency physician to provide medical clearance. The behavioral health service begins their psychiatric evaluation of the patient simultaneously with the medical clearance process. The behavioral health evaluation will determine the need for psychiatric admission together with the emergency service.

The emergency service is responsible for the evaluation and treatment of a patients' agitation. A treatment protocol with a scale of agitation is used to guide the physician into whether to restrain or medicate a patient as well as the type and dosage of medication.

A convenience sample of patients who present with psychiatric complaints to the emergency department when a research fellow from the Department of Emergency Medicine is available will be enrolled in the study.

Inclusion/Exclusion Criteria

Patients can be enrolled in the study only if they meet all of the following criteria:

1. Presenting with a psychiatric complaint.
2. Male or female patients at least 18 years of age.
3. Patients must be emergency department patients during the study.
4. Each patient, or a patient's legal representative (as allowed by local law), must understand the nature of the study and must agree to study enrollment.
5. English speaking.
6. Consenting

Patients will be excluded from the study for any of the following reasons:

1. Unstable patients
2. Patients who have delirium or dementia will be excluded because of its complicated medical rather than psychiatric etiologies.
3. Prisoners
4. Pediatric patients The research fellow will obtain consent from the patient or their surrogate and ensure that the patient meets all study inclusion and no exclusion criteria. The researcher will provide a brief overview of the study to the patient to obtain verbal consent.

Information will be collected on a data collection sheet that will include basic demographic information on the patient: age, gender, diagnosis, current medication, restraint usage, time restraints were applied and type, dose and time medication is administered. A research fellow will complete the data collection sheet and input the data of enrolled patients into a database. The statistician will perform an analysis of the data looking for statistical significance of the data to the posed questions. Once all data is collected, any identifying information on the patient will be destroyed to ensure patient confidentiality.

The research fellow will be responsible for completing an agitation checklist on each patient enrolled in the study. The patients' psychiatric diagnosis will be noted from the psychiatric service.

The patients were evaluated for their level of agitation at arrival and every 30 minutes for 2 hours. We will use four tests of agitation: Brief Agitation Tool, Positive and Negative Syndrome Scale-Excited Component, Agitation Behavior Scale, and the Psychological Pain Assessment Scale.The independent variables will be diagnosis, number of restraints administered (if any), time intervals every 30 minutes of each test, type of medication administered ( if any), and time to non-agitated state level on each scale. The dependent variables would be the assessing psychic pain using the level of agitation as a surrogate marker.

The data will be inputted into a Statistical Program for Social Science program for analysis. Group differences between cases and levels of agitation will be examined by two-tailed t-tests and analysis of variance. Analysis of variance and its derivatives will be used to determine what, if any, differences exist between the patient's agitation and psychological pain scale assessments at 30 minute intervals up to the two hour mark. Because the relation between the predictor and outcome variables is not presumed to be a linear function, the measure of association between the outcome of interest and the predictor variable is represented by an odds ratio instead of a multiplicative factor. Comparisons of odds ratio between predictor variables help determine the factors of greatest importance, while their confidence intervals will indicate their statistical significance. This will determine the probability of which test will accurately predict the lowering levels of agitation at timed intervals as compared to each other and to the dependent variable. Additionally, it can predict any correlations to the independent variables which may influence the outcomes such as gender, age and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Patients can be enrolled in the study only if they meet all of the following criteria:

1. Presenting with a psychiatric complaint.
2. Male or female patients at least 18 years of age.
3. Patients must be emergency department patients during the study.
4. Each patient, or a patient's legal representative (as allowed by local law), must understand the nature of the study and must agree to study enrollment.
5. English speaking.
6. Consenting

Exclusion Criteria:

1. Unstable patients
2. Patients who have delirium or dementia will be excluded because of its complicated medical rather than psychiatric etiologies.
3. Prisoners
4. Pediatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of patients who presented with psychiatric complaints to the emergency department when a research fellow from the Department of Emergency Medicine is available in the ED will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Brief Agitation Measure | 5 MINUTES
  The Brief Agitation Measure is a three question tool: (1) I want to crawl out of my skin,(2) I feel so stirred up inside I want to scream and (3) I feel a lot of emotional turmoil in my gut. Each item is scored from 1-7 so the scores are from 3-21. Higher scores are considered great level of agitation.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale | 3 hours
  The Positive and Negative Syndrome Scale is a commonly used instrument, to assess severely aggressive and agitated patients. The tool consists of 5 items: excitement, tension, hostility, being uncooperative, and poor impulse control.
  The 5 items are rated from 1 (not present) to 7 (extremely severe); scores range from 5 to 35; mean scores ≥ 20 clinically correspond to severe agitation.

OTHER OUTCOMES:
Agitation Calmness Evaluation Scale | 15-20 minutes
  Semi structured interview with patients
Psychological Pain Assessment Scale | 3 hours
  The Psychological Pain Assessment Scale was designed to fill the need for a brief, easily understood instrument to assess both frequency and intensity of psychological pain.

CONTACTS AND LOCATIONS:
Overall Officials: Les Zun, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be available to other researchers. Data will only be shared through publications and presentations once the study has been completed.

REFERENCES:
- [Background] Shneidman ES. The psychological pain assessment scale. Suicide Life Threat Behav. 1999 Winter;29(4):287-94. No abstract available. PMID 10636323
- [Background] Mee S, Bunney BG, Bunney WE, Hetrick W, Potkin SG, Reist C. Assessment of psychological pain in major depressive episodes. J Psychiatr Res. 2011 Nov;45(11):1504-10. doi: 10.1016/j.jpsychires.2011.06.011. Epub 2011 Aug 9. PMID 21831397
- [Background] Shattell MM. Why does "pain management" exclude psychic pain? Issues Ment Health Nurs. 2009 May;30(5):344. doi: 10.1080/01612840902844890. No abstract available. PMID 19437255
- [Background] Flor H. Psychological pain interventions and neurophysiology: implications for a mechanism-based approach. Am Psychol. 2014 Feb-Mar;69(2):188-96. doi: 10.1037/a0035254. PMID 24547804